CLINICAL TRIAL: NCT03698305
Title: A Double-blinded, Randomized, Controlled, Single Ascending Dose Study in Healthy Adult Volunteers to Assess the Safety and Pharmacokinetics of an Investigational Imaging Product
Brief Title: A Study in Healthy Adult Volunteers to Assess the Safety and Pharmacokinetics of an Investigational Imaging Product
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5354-CL-0001
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2020-04

CONDITIONS: Healthy Subjects
Keywords: Tolerability; Pharmacokinetics; Safety; ASP5354

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ASP5354 Dose Escalation (5 Dose Levels) (Experimental): Healthy male and female subjects will be assigned to Cohorts 1-5. In each cohort, 4 subjects will be randomized to receive escalated doses of ASP5354. Each subject will receive a single intravenous bolus injection under fasting conditions.
  Interventions: Drug: ASP5354
- Placebo Dose Escalation (5 Dose Levels) (Placebo Comparator): Healthy male and female subjects will be assigned to Cohorts 1-5. In each cohort, two subjects will be randomized to receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP5354 — Intravenous
  Arms: ASP5354 Dose Escalation (5 Dose Levels)
Drug: Placebo — Intravenous
  Arms: Placebo Dose Escalation (5 Dose Levels)

SUMMARY:
The objective of this study is to assess the safety and tolerability of ASP5354 administered intravenously as a single dose to healthy subjects. This study will also assess the single dose pharmacokinetics of ASP5354 in plasma and urine.

DETAILED DESCRIPTION:
This is a study comprising of 5 cohorts (cohorts 1 to 5) of 6 healthy subjects in each cohort (4 in each ASP5354 cohort and 2 in each placebo cohort). If the data from cohorts 1 to 3 are sufficient to characterize safety, tolerability and pharmacokinetics and the assessed doses reach the expected urine ASP5354 concentration, the study may be ended without running the fourth or fifth cohorts.

ELIGIBILITY:
Inclusion Criteria:

* A female subject is eligible to participate if she is not pregnant and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP). OR
  * A WOCBP who agrees to follow the contraceptive guidance throughout the treatment period and for at least 30 days after the final investigational product (IP) administration.
* Female subject must agree not to breastfeed starting at screening, throughout the study period and for 30 days after the final IP administration.
* Female subject must not donate ova starting at screening, throughout the study period and for 30 days after the final IP administration.
* Male subject with female partner(s) of childbearing potential must agree to use contraception during the treatment period and for at least 30 days after the final IP administration.
* Male subject must not donate sperm during the treatment period and for at least 30 days after the final IP administration.
* Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom with spermicide for the duration of the pregnancy or time the partner is breastfeeding throughout the study period and for 30 days after the final IP administration.
* Subject agrees not to participate in another interventional study while participating in the present study.
* Subject has a body mass index range of 18.5 to 32.0 kg/m2, inclusive, and weighs > 50 kg (for males) or > 40 kg (for females) at screening.

Exclusion Criteria:

* Subject has signs of urinary tract infection, abnormalities or disease or has had operational interventions on the urinary tract.
* Subject has received any IP within 28 days or 5 half-lives (if known), whichever is longer, prior to screening.
* Female subject who has been pregnant within 6 months prior to screening or breastfeeding within 3 months prior to screening.
* Subject has a known or suspected hypersensitivity to ASP5354 or any components of the formulation used.
* Subject has had previous exposure to ASP5354.
* Subject has any of the liver function tests (aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase, gamma glutamyl transferase and total bilirubin [TBL]) > upper limit of normal (ULN) at day -1.
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies) prior to IP administration.
* Subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy.
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection) or fungal (noncutaneous) infection within 2 weeks prior to day -1.
* Subject has any clinically significant abnormality following the physical examination, electrocardiogram (ECG) and protocol-defined clinical laboratory tests at screening or day 1.
* Subject has a mean pulse < 45 bpm or > 90 bpm, mean systolic blood pressure > 140 mmHg or mean diastolic blood pressure > 90 mmHg at day -1.
* Subject has a mean corrected QT interval using Fridericia's formula (QTcF) > 430 msec (for males) and > 450 msec (for females) at day 1 (as determined by the ECG machine). If the mean QTcF exceeds the limits above, 1 additional triplicate (3 measurements) ECG can be taken.
* Subject has used any prescribed or nonprescribed drugs (including vitamins, oral contraceptives, hormone replacement therapy or natural and herbal remedies [e.g., St. John's Wort]) in the 2 weeks prior to IP administration, except for occasional use of acetaminophen (up to 2 g/day) or topical dermatological products, including corticosteroid products.
* Subject has smoked or has used tobacco-containing products or nicotine or nicotine containing products in the past 6 months prior to screening or the subject tests positive for cotinine at screening or day -1.
* Subject has a history of consuming more than 14 units of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical/substance abuse within the past 2 years prior to screening (Note: 1 unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits/hard liquor).
* Subject has used any drugs of abuse (including but not limited to amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and opiates) within 3 months prior to day -1 or the subject tests positive for alcohol or drugs of abuse (including but not limited to amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and opiates) at screening or day -1.
* Subject has used any inducer of metabolism (e.g., barbiturates and rifampin) in the 3 months prior to day -1.
* Subject has had significant blood loss, donated 1 unit (450 mL) or more of blood or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to day -1.
* Subject has a positive serology test for hepatitis B surface antigen, hepatitis B core antibody, hepatitis A virus antibodies (immunoglobulin M), hepatitis C virus antibodies or human immunodeficiency virus p24 antigen at screening.
* Subject has any of the renal function tests (blood urea nitrogen and creatinine) > ULN at day -1.

In such a case, the assessment may be repeated once.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessed by nature, frequency, and severity of Adverse Events (AEs) | Up to Day 14
  An AE is any untoward medical occurrence in a participants administered ASP5354, and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of a medicinal product whether or not considered related to the medicinal product.
  AEs will be coded using MedDRA.
Number of participants with laboratory value abnormalities and/or AEs | Up to Day 7
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and /or AEs | Up to Day 7
  Number of participants with potentially clinically significant vital sign values.
Safety and tolerability assessed by 12-lead electrocardiogram (ECG) | Up to Day 7
  12-lead ECGs will be taken after the subject has been resting in the supine position for at least 5 minutes. 12 lead ECGs will be taken in triplicate.
Number of participants with physical exam abnormalities and/or adverse events (AEs) | Up to Day 7
  Number of participants with potentially clinically significant physical exam values.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ASP5354 in plasma: plasma concentration at time 0 (C0) | Before dosing on Day 1
  C0 will be derived from the PK samples collected.
PK of ASP5354 in plasma: area under the concentration-time curve from time zero to 24 hours postdose (AUC0-24) | Up to 24 hr after dosing
  AUC0-24 will be derived from the PK samples collected.
PK of ASP5354 in plasma: AUC extrapolated from time to infinity as a percentage of total area under the concentration-time curve (AUCinf) | Up to 24 hr after dosing
  AUCinf will be derived from the PK samples collected.
PK of ASP5354 in plasma: AUC from time zero to the time of the last quantifiable concentration (AUClast) | Up to 24 hr after dosing
  AUClast will be derived from the PK samples collected.
PK of ASP5354 in plasma: AUC extrapolated from time to infinity as a percentage of total area under the concentration-time curve (AUCinf(%extrap)) | Up to 24 hr after dosing
  AUCinf (%extrap) will be derived from the PK samples collected.
PK of ASP5354 in plasma: maximum concentration (Cmax) | Up to 24 hr after dosing
  Cmax will be derived from the PK samples collected.
PK of ASP5354 in plasma: total body clearance of drug from plasma (CL) | Up to 24 hr after dosing
  CL will be derived from the PK samples collected.
PK of ASP5354 in plasma: time of maximum concentration (tmax) | Up to 24 hr after dosing
  tmax will be derived from the PK samples collected.
PK of ASP5354 in plasma: apparent terminal elimination half-life (t1/2) | Up to 24 hr after dosing
  t1/2 will be derived from the PK samples collected.
PK of ASP5354 in plasma: volume of distribution during terminal phase (Vz) | Up to 24 hr after dosing
  Vz will be derived from the PK samples collected.
PK of ASP5354 in urine: amount of unchanged drug excreted into the urine (Ae) | Up to 24 hr after dosing
  Ae will be derived from the PK samples collected.
PK of ASP5354 in urine: percentage of dose excreted in the urine (Ae%) | Up to 24 hr after dosing
  Ae% will be derived from the PK samples collected.
PK of ASP5354 in urine: cumulative amount of unchanged drug excreted into the urine (CumAe) | Up to 24 hr after dosing
  CumAe will be derived from the PK samples collected.
PK of ASP5354 in urine: cumulative percentage of dose excreted in the urine (CumAe%) | Up to 24 hr after dosing
  CumAe% will be derived from the PK samples collected.
PK of ASP5354 in urine: amount of unchanged drug excreted into the urine from time zero to the time of the last quantifiable concentration (Aelast) | Up to 24 hr after dosing
  Aelast will be derived from the PK samples collected.
PK of ASP5354 in urine: percent of unchanged drug excreted into the urine from time zero to the time of the last quantifiable concentration (Aelast%) | Up to 24 hr after dosing
  Aelast% will be derived from the PK samples collected.
PK of ASP5354 in urine: renal clearance (CLR) | Up to 24 hr after dosing
  CLR will be derived from the PK samples collected.
PK of ASP5354 in urine: mean ASP5354 urine concentrations at each time point | Up to 24 hr after dosing
  Mean ASP5354 urine concentrations will be derived from the PK samples collected.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- Covance CRU, Daytona Beach, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.